CLINICAL TRIAL: NCT00478439
Title: Investigation of Macular Pigment Augmentation on Dark Adaptation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated: Recruitment delay due to equipment malfunction
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: ZeaVision, Inc. (Industry)
Responsible Party: Leo P. Semes, O.D./Principal Investigator, UAB School of Optometry
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: F070410002
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Aging; Age-Related Macular Degeneration
Keywords: aging; age-related macular degeneration; macular pigment; dark adaptation
MeSH Terms: conditions — Macular Degeneration | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo Comparator (Placebo Comparator)
  Interventions: Dietary Supplement: ZeaVision EyePromise Restore; Dietary Supplement: Multivitamin

INTERVENTIONS:
Dietary Supplement: ZeaVision EyePromise Restore — Vitamin C 120mg, Vitamin E 60IU, Zinc 15mg, Fish Oil 250mg, Omega 3 125mg, Alphaliploic acid 10mg, Zeaxanthin 8mg,mixed tocopherols 6mg, lutein 4mg,
Dietary Supplement: Multivitamin — Vitamin C 120mg, Vitamin E 60IU, Zinc 15mg, Fish Oil 250mg, Omega 3 125mg, Alphaliploic acid 10mg, mixed tocopherols 6mg, lutein 4mg,

SUMMARY:
The study will evaluate whether taking a nutritional supplement designed to increase macular pigment in the eye can improve a person's ability to adjust to darkness. Patients will be assigned to take either a placebo or nutritional supplement for 8 months. Vision will be assessed at baseline, 4 months, and 8 months.

DETAILED DESCRIPTION:
The study design is a randomized, double-blinded, placebo-controlled intervention study that will evaluate whether macular pigment augmentation improves the speed of dark adaptation. Two groups of participants will be enrolled, old adults with normal vision and early age-related macular degeneration patients. Macular pigment will be augmented using EyePromise RESTORE (ZeaVision, Inc). EyePromise RESTORE is a nutritional supplement that has been found to increase macular pigment levels in some users. Macular pigment level and the speed of dark adaptation (how fast a person adjusts to the dark) will be assessed at baseline, 4-months, and 8-months. Fundus appearance will be assessed at baseline and 8-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 80 years old
* < +- 4.00 diopters spherical equivalent
* normal eye health or early age-related macular degeneration

Exclusion Criteria:

* neurological conditions that can impair vision
* diabetes

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Dark Adaptation | Measured 3 times over 8 months

SECONDARY OUTCOMES:
Macular Pigment Density | Measured 3 times over 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Leo P Semes, O.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB School of Optometry, Birmingham, Alabama, United States